CLINICAL TRIAL: NCT01025596
Title: A PHASE I/IIa DOSE ESCALATION STUDY IN ASIA OF REPEATED ADMINISTRATION OF "CYT107" (Glyco-r-hIL-7) ADDED ON TREATMENT IN GENOTYPE 1 HCV INFECTED PATIENTS RESISTANT TO PEGYLATED INTERFERON-ALPHA AND RIBAVIRIN
Brief Title: Dose Escalation Study of IL-7 and Bi-therapy in HCV Patients Resistant After 12 Weeks of Bi-therapy (ECLIPSE 1)
Acronym: ECLIPSE 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-05; EudraCT number 2006-006024-20
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: interleukin-7; immune-based therapies; hepatitis C; chronic hepatitis; resistance to Peg-interferon and ribavirin bi-therapy; immune specific responses to HCV; phase 1; viral disease; liver disease
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic; Virus Diseases; Liver Diseases | interventions — Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYT107 (Experimental)
  Interventions: Drug: Interleukin-7

INTERVENTIONS:
Drug: Interleukin-7 — 4dose levels: 3, 10, 20 and 30µg/kg. 4 administrations, 1 per week

SUMMARY:
This study will evaluate the safety of a new experimental drug, IL-7, in people with HCV infection resistant after 12 weeks of bi-therapy.

DETAILED DESCRIPTION:
This is a Phase I inter-patient dose-escalation study assessing weekly doses of Interleukin-7 (CYT107) in adult patients infected by Genotype 1 Virus of Hepatitis C and resistant to standard treatment with Peg-Interferon and Ribavirin (biotherapy)after 12 weeks of this standard bi-therapy.

The dose escalation is aimed at establishing the safety of a biologically active doses of CYT107 added to the combination therapy of pegylated interferon-alpha and ribavirin. At each dose level, study patients will receive a subcutaneous administration of CYT107 per week for a total of 4 administrations.

Groups of 3 to 6 patients will be entered at each dose level of CYT107. Four dose levels are planned.

Eligible patients will a cycle of four weekly injections at a defined dose level in addition to the bi-therapy. Standard bi-therapy will continue 4 weeks after CYT107 treatment discontinuation. The duration of study is approximately 11 weeks including screening period.

Participants have 1 hospitalization overnight and 8 clinic visits. The four administrations are sub-cutaneous and are given as a shot under the skin in the arm or abdomen or leg.

During the study visits the following may be done:

* Medical history, physical examination, blood tests every visit.
* Electrocardiogram (EKG)
* Chest x-ray study
* Liver/spleen imaging
* Blood sample collections at frequent intervals
* Urine tests several times during the study.

ELIGIBILITY:
Main Inclusion Criteria:

* Genotype I infected patients
* Age > 18 years
* Absence of early viral response to a first treatment with PEG-interferon-alpha plus ribavirin given for at least 12 weeks. Absence of early viral response (EVR) will be defined as detectable HCV with a decrease HCV RNA load < 2 logs, measured by a quantitative PCR tests, as compared to baseline levels measured by a similar technique
* Ongoing treatment by PEG-interferon-alpha plus ribavirin at study entry

Main Exclusion Criteria:

* Infection by HBV
* Infection by HIV-1 and /or HIV-2
* Apart from HCV infection, presence of active infection requiring a specific treatment or a hospitalization
* Cirrhosis (Metavir F4) assessed by biopsy or FibroScan® or by liver biopsy within the last 6 months prior CYT107 treatment initiation. If assessed by Fibroscan® patients with a result > 10 KPa will be excluded
* Other liver disease (notably from alcoholic, metabolic or immunological origin)
* Body mass index (BMI) > 30kg/m2
* Inability to give informed consent
* Administration of growth factors (G-CSF, EPO) within the 12 weeks of the combination therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety of biologically active doses of CYT107 added to a standard bi-therapy in patients with a chronic infection by a genotype 1 Hepatitis C Virus (HCV) not responding to this combination therapy 12 weeks after its initiation. | 8 weeks after start of CYT107

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics of CYT107 in this patients population. | As primary
potential anti-viral effect of CYT107 | As primary
immune specific response to HCV | As primary

CONTACTS AND LOCATIONS:
Overall Officials: Tilman Gerlach, Study Chair — University of Zurich / Saint Gallen
Locations (7):
- France (4):
  - Hopital Jean Verdier, Bondy
  - Beaujon Hospital, Clichy
  - Hopital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hopital Civil, Strasbourg
- Italy (2):
  - Azienda Ospedaliero-Universitaria, Policlinico Sant'Orsola Malpighi, Bologna
  - San Raffaele Scientific Institute, Milan
- University of Zurich, Zurich, Switzerland